CLINICAL TRIAL: NCT04019444
Title: A Phase 1, Dosage-Escalation Study of the Safety and Immunogenicity of a Novel Rabies Vaccine ChAd155-RG vs. the Comparator RABAVERT Vaccine in Healthy Adult Subjects
Brief Title: Dosage-Escalation Study of the Safety and Immunogenicity of a Novel Rabies Vaccine ChAd155-RG vs. the Comparator RABAVERT Vaccine in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 17-0089
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2019-07-05

CONDITIONS: Rabies; Rabies Immunisation
Keywords: Adults; ChAd155-RG; Dosage-Escalation; Healthy; Immunogenicity; RABAVERT; Rabies; Safety; Vaccine
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A (Experimental): One dose (1 ml (5x10^10 vp)) of ChAd155-RG vaccine administered intramuscularly on Day 1, and 1 ml of matching placebo administered intramuscularly on Days 8, 15, 22. N=14 (3 sentinel, 11 non-sentinel)
  Interventions: Biological: ChAd155-RG; Other: Placebo
- Arm B (Experimental): One dose (1 ml (1x10^11 vp)) of ChAd155-RG vaccine administered intramuscularly on Day 1, and 1 ml of matching placebo administered intramuscularly on Days 8, 15, 22. N=14 (3 sentinel, 11 non-sentinel)
  Interventions: Biological: ChAd155-RG; Other: Placebo
- Arm C (Experimental): Two doses (1 ml (1x10^11 vp) each) of ChAd155-RG vaccine administered intramuscularly on Day 1 (first dose) and Day 15 (second dose), and 1 ml of matching placebo administered intramuscularly on Days 8 and 22. N=10
  Interventions: Biological: ChAd155-RG; Other: Placebo
- Arm D (Active Comparator): Three doses (1 ml each) of RABAVERT vaccine administered intramuscularly on Day 1 (first dose), Day 8 (second dose), and Day 22 (third dose), and 1 ml of matching placebo administered intramuscularly on Day 15. N=12 (2 sentinel, 10 non-sentinel)
  Interventions: Other: Placebo; Biological: Rabies Vaccine

INTERVENTIONS:
Biological: ChAd155-RG — The ChAd155-RG Vaccine consists of a replication-defective group C ChAd, ChAd155, expressing RG under the control of the CMV promoter. The RG sequence cloned into the ChAd155 vector is a medoid, a natural viral strain with the highest average percent of amino acid identity among all RG sequences annotated in the NCBI database. The selected RG (NCBI strain AGN94271) shares an average 94% percent identity to the RGs in current vaccines.
  Arms: Arm A; Arm B; Arm C
Other: Placebo — 0.9% Sodium Chloride, USP injection.
Biological: Rabies Vaccine — The RABAVERT Vaccine is an inactivated, purified chick embryo cell vaccine (PCECV). It consists of lyophilized rabies virus (strain Flury LEP) that has been propagated in chicken fibroblasts, inactivated with beta-propiolactone, and concentrated and purified by centrifugation
  Arms: Arm D

SUMMARY:
This is a single-center, observer-blinded, dosage-escalation trial to evaluate the safety, tolerability, reactogenicity, and immunogenicity of ChAd155-RG compared with RABAVERT in rabies virus-naïve healthy male and non-pregnant female adult subjects ages 18-49. There are 4 dose groups: Group A will receive ChAd155-RG at the lower dosage (5x1010vp) on Day 1, then placebo injections on Days 8, 15, and 22; Group B will receive ChAd155-RG at the higher dosage (1x1011vp) on Day 1, then placebo injections on Days 8, 15, and 22; Group C will receive ChAd155-RG at the higher dosage (1x1011vp) on Days 1 and 15, and placebo injections on Days 8 and 22; Group D will receive RABAVERT at the standard dose (1 mL) on Days 1, 8, and 22, and a placebo injection on Day 15. Since this is a dosage-escalation study, sentinel subjects will be used at each dosage level before non-sentinel subjects will be enrolled. The study will be conducted at Emory University Vaccine and Treatment Evaluation Unit (VTEU). This trial is expected to take approximately 48 months to complete. The duration of each subject's participation is approximately 13 months, from recruitment through the last study visit. The primary objectives of this study are: 1) Assessment of the safety, tolerability, and reactogenicity of one dose of ChAd155-RG at 5x1010vp per dose, or one or two doses of ChAd155-RG at 1x1011vp per dose; 2) Comparison of the safety, tolerability, and reactogenicity of one or two doses of ChAd155-RG, with three doses of RABAVERT.

DETAILED DESCRIPTION:
This is a single-center, observer-blinded, Phase 1, dosage-escalation trial to evaluate the safety, tolerability, reactogenicity, and immunogenicity of ChAd155-RG compared with RABAVERT in rabies virus-naïve healthy male and non-pregnant female adult subjects ages 18-49. Subjects who have never received a licensed or investigational rabies virus vaccine, or an Ad-based investigational vaccine, and who have never been exposed to a rabid animal will be eligible for enrollment. There are 4 dose groups: Group A will receive ChAd155-RG at the lower dosage (5x1010vp) on Day 1, then placebo injections on Days 8, 15, and 22; Group B will receive ChAd155-RG at the higher dosage (1x1011vp) on Day 1, then placebo injections on Days 8, 15, and 22; Group C will receive ChAd155-RG at the higher dosage (1x1011vp) on Days 1 and 15, and placebo injections on Days 8 and 22; Group D will receive RABAVERT at the standard dose (1 mL) on Days 1, 8, and 22, and a placebo injection on Day 15. Since this is a dosage-escalation study, sentinel subjects will be used at each dosage level before non-sentinel subjects will be enrolled. The SMC will review the available safety, reactogenicity, AE, and lab data of all the sentinel subjects, and will decide if the remaining non-sentinel subjects should be enrolled. The study will be conducted at Emory University Vaccine and Treatment Evaluation Unit (VTEU). This trial is expected to take approximately 48 months to complete. The duration of each subject's participation is approximately 13 months, from recruitment through the last study visit. The primary objectives of this study are: 1) Assessment of the safety, tolerability, and reactogenicity of one dose of ChAd155-RG at 5x1010vp per dose, or one or two doses of ChAd155-RG at 1x1011vp per dose; 2) Comparison of the safety, tolerability, and reactogenicity of one or two doses of ChAd155-RG, with three doses of RABAVERT. The secondary objective is to assess the serum rabies VNA levels by a standard, WHO-approved, RFFIT, as assessed by immune response kinetics (through approximately 12 months after first dose of vaccine), seroconversion rates, and peak GMT in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a male or female aged 18-49 years old (inclusive) at the time of first vaccination.
2. Must be able to provide written informed consent.
3. Must have a body mass index (BMI) = / >18.5 and <35.0 kg/m^2
4. Must be in good health based on physical examination, vital signs*, medical history, safety labs**, and the investigator's clinical judgment.

   *Vital signs must be within the normal ranges. If a subject has elevated systolic or diastolic blood pressure, subject may rest for 10 minutes in a quiet room and the blood pressure may be retaken.

   **Safety lab normal ranges will be those used by the reference clinical lab. Protocol-specific criteria for individual subjects are listed in criteria #5.
5. Must have acceptable* lab values within 28 days before enrollment. *Acceptable values include:

   * Hemoglobin: women >11.6 g/dL, men >13.1 g/dL
   * White blood cells: >3,700 but <10,900 cells/mm^3
   * Absolute neutrophil count: = / >1,500 cells/mm^3
   * Absolute lymphocyte count: = / >850 cells/mm^3
   * Platelets: >139,000 but <401,000 per mm^3
   * Urine dipstick (clean urine sample): protein <1+, glucose negative
   * Alanine transaminase and aspartate transaminase (ALT, AST) <1.1 x institutional upper limit of normal (ULN)
   * Total bilirubin <1.1x institutional ULN
   * Blood urea nitrogen (BUN) <1 x institutional ULN
   * Serum creatinine <1x institutional ULN
   * If lab screening tests are out of range, repeating them is permitted once, provided there is an alternative explanation for the out-of-range value.
6. Women of childbearing potential* must have a negative serum pregnancy test at screening and negative urine pregnancy tests within 24 hours before each vaccination.

   * Women of non-childbearing potential, defined as postmenopausal (any age with amenorrhea for = / >12 months without other known or suspected cause for amenorrhea), or surgically sterile [hysterectomy, bilateral tubal ligation, bilateral oophorectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization)] with documented confirmation test = / >3 months after the procedure), are not required to use contraceptive methods.
7. Women of childbearing potential must use an acceptable method of contraception* from 28 days before the first vaccination until = / >60 days after the last vaccination.

   *Acceptable methods of contraception include: prescription oral contraceptives, contraceptive injections, intrauterine device (IUD), implants, vaginal ring, double-barrier method, contraceptive patch, male partner who had a vasectomy at least 6 months prior to study enrollment, abstinence (defined as refraining from heterosexual intercourse during participation in this trial [from 28 days before the first vaccination until = / >60 days after the last vaccination]).
8. Female subjects must agree to not donate eggs (ova, oocytes) from the start of screening until = / >60 days after the last vaccination.
9. Male subjects who have not had a vasectomy* and are sexually active with a woman of childbearing potential must agree to use an acceptable method of contraception**.

   *Men who have had a vasectomy must have had the procedure performed at least 6 months prior to study enrollment.

   **Acceptable methods of contraception must be used from the first vaccination until = / >60 days after the last vaccination, and include: abstinence (defined as refraining from heterosexual intercourse with a female partner of childbearing potential during participation in this trial [from 28 days before the first vaccination until = / >60 days after the last vaccination]; a double-barrier method, such as condom with spermicidal foam/gel/film/cream/suppository and partner with occlusive cap (diaphragm, cervical/vault caps); if the female partner is using an acceptable method of contraception (see Inclusion Criterion #7), a single-barrier method for the male subject is acceptable.
10. Male subjects must agree to not donate sperm from the start of screening until = / >60 days after the last vaccination.
11. Must be available and willing to participate for the duration of this trial.
12. Must have a means to be contacted by telephone.

Exclusion Criteria:

1. Was ever vaccinated with a licensed or investigational rabies vaccine* or was diagnosed with rabies exposure, infection, or disease.

   *Includes RABAVERT and Imovax. Subject's verbal history will suffice.
2. Has a higher risk than the average US resident with regard to exposure to rabies, per the Rabavert package insert and rabies vaccination recommendations from the CDC*.

   * People at high risk of exposure to rabies, such as veterinarians, animal handlers, rabies laboratory workers, spelunkers, and rabies biologics production workers.
   * People whose activities bring them into frequent contact with rabies virus or with possibly rabid animals.
   * International travelers who are likely to come in contact with animals in parts of the world where rabies is common.
3. Was ever vaccinated with a licensed or investigational Ad vector or Ad vaccine.
4. Is currently taking chloroquine or hydroxychloroquine.
5. Was diagnosed with laboratory-confirmed COVID-19 (PCR or antigen-based test) in the preceding 28 days.
6. Positive serology for HIV antibody, HCV antibody, or Hepatitis B surface antigen (HBsAg).
7. Has known allergy or history of anaphylaxis or other serious adverse reaction to a vaccine or vaccine products*.

   *Including egg products, aminoglycosides, gelatin, sorbitol, tris (hydroxymethyl)-amino methane (THAM), or any of the constituents of the study vaccines.
8. Has severe allergy or anaphylaxis to latex.
9. Has an acute illness or temperature = / >38.0 Degrees Celsius on Day 1*.

   *Subjects with fever or acute illness on the day of vaccination may be re-assessed and enrolled if healthy or only minor residual symptoms remain within 3 days.
10. Female subjects who are pregnant or breastfeeding, or planning to become pregnant while enrolled in this trial and at least 60 days after last vaccination.
11. Has history of autoimmune disease, or clinically significant cardiac, pulmonary, hepatic, rheumatologic, or renal disease by history, physical examination, and/or lab studies.
12. Has history of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure*.

    *Subjects with a history of skin cancer must not be vaccinated at the previous tumor site.
13. Has known or suspected congenital or acquired immunodeficiency, or recent history or current use of immunosuppressive therapy*.

    *Anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term (= / >2 weeks within the previous 3 months) systemic corticosteroid therapy (at a dosage of = / >0.5 mg/kg/day). Intranasal or topical prednisone (or equivalent) are allowed.
14. Is post-organ and/or stem cell transplant, whether or not on chronic immunosuppressive therapy.
15. Had major surgery (per the investigator's judgment) within 4 weeks before study entry or planned major surgery during this trial.
16. Has history of diabetes mellitus type 1 or type 2, including cases controlled with diet alone.

    *Note: history of isolated gestational diabetes is not an exclusion criterion.
17. Has history of thyroidectomy, or thyroid disease requiring medication in the last 12 months.
18. Has history of hypertension, even if medically controlled.

    *Note: Vital signs must be normal by protocol toxicity grading scale. In the event of an abnormal heart rate or blood pressure due to physiological variation or activity, the subject may rest for 10 minutes in a quiet room, and then blood pressure and/or heart rate re-measured. Repeated vital signs may be used to determine eligibility.
19. Received live attenuated vaccines from 30 days before first vaccination until 30 days after final vaccination*.

    *Not including licensed or authorized COVID-19 vaccines.
20. Received killed or inactivated vaccines from 14 days before first vaccination until 30 days after final vaccination*.

    *Not including licensed COVID-19 vaccines
21. Received experimental therapeutic agents within 3 months before first vaccination or plans to receive any experimental therapeutic agents during this trial*.

    *That that in the opinion of the investigator would interfere with safety or immunogenicity assessments.
22. Is currently participating or plans to participate in another clinical study which would involve receipt of the following:*

    * An investigational product, blood drawing, or an invasive medical procedure that would require administration of anesthetics, intravenous (IV) dyes, or removal of tissue during this trial and, in the opinion of the investigator, would interfere with safety or immunogenicity assessments.

    -Includes endoscopy, bronchoscopy, and administration of IV contrast.
23. Received blood products or immunoglobulin in the 3 months before study entry or planned use during this trial.
24. Donated a unit of blood or blood products within 8 weeks before Day 1 or plans to donate blood or blood products during this trial.
25. Has major psychiatric illness in the past 12 months that in the opinion of the investigator would preclude participation.
26. Has current alcohol use or current or past abuse of recreational or narcotic drugs by history as judged by the investigator to potentially interfere with study adherence.
27. Has a history of chronic urticaria.
28. Has tattoos, scars, or other marks on both deltoid areas which would, in the opinion of the investigator, interfere with assessment of the vaccination site.
29. Is a site employee* or staff who are paid entirely or partially by/through the OCRR contract for this trial, or staff who are supervised by the Principal Investigator (PI) or sub-investigators.

    *Including the PI, sub-investigators listed on Form FDA 1572 or Investigator of Record Form.
30. In the opinion of the investigator cannot communicate reliably, is unlikely to adhere to the requirements of this trial, or has any condition which would limit the ability to complete this trial.
31. Has history of Guillain-Barre syndrome, meningitis, encephalitis, neuroparalysis, transient paralysis, myelitis, retrobulbar neuritis, multiple sclerosis, vertigo, or visual disturbances.
32. Has a history of arterial or venous thrombosis, or thrombocytopenia that required medical attention.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hope Clinic of Emory University, Decatur, Georgia, United States

REFERENCES:
- [Derived] Phadke VK, Gromer DJ, Rebolledo PA, Graciaa DS, Wiley Z, Sherman AC, Scherer EM, Leary M, Girmay T, McCullough MP, Min JY, Capone S, Sommella A, Vitelli A, Retallick J, Seetahal J, Koller M, Tsong R, Neill-Gubitz H, Mulligan MJ, Rouphael NG. Safety and immunogenicity of a ChAd155-vectored rabies vaccine compared with inactivated, purified chick embryo cell rabies vaccine in healthy adults. Vaccine. 2024 Dec 2;42(26):126441. doi: 10.1016/j.vaccine.2024.126441. Epub 2024 Oct 16. PMID 39418686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy adult volunteers meeting all protocol-defined eligibility criteria. Participants were recruited through IRB-approved flyers on the Emory University campus, social media, list serves, clinical trial recruitment websites, a HIPAA-compliant clinical trials database to identify participants of previous trials at the Hope Clinic who had agreed to future contact, presentations by Hope Clinic faculty, and word-of-mouth. Enrollment occurred between 19SEP2019 and 07MAR2022.
Groups:
- Low Dose ChAd155-RG: One dose (1 ml (5x10^10 vp)) of ChAd155-RG vaccine administered intramuscularly on Day 1, and 1 ml of matching placebo administered intramuscularly on Days 8, 15, and 22.
- High Dose ChAd155-RG (x1): One dose (1 ml (1x10^11 vp)) of ChAd155-RG vaccine administered intramuscularly on Day 1, and 1 ml of matching placebo administered intramuscularly on Days 8, 15, and 22.
- High Dose ChAd155-RG (x2): Two doses (1 ml (1x10^11 vp) each) of ChAd155-RG vaccine administered intramuscularly on Day 1 (first dose) and Day 15 (second dose), and 1 ml of matching placebo administered intramuscularly on Days 8 and 22.
- RABAVERT: Three doses (1 ml each) of RABAVERT vaccine administered intramuscularly on Day 1 (first dose), Day 8 (second dose), and Day 22 (third dose), and 1 ml of matching placebo administered intramuscularly on Day 15.
Period: Overall Study
Arm/Group | Low Dose ChAd155-RG | High Dose ChAd155-RG (x1) | High Dose ChAd155-RG (x2) | RABAVERT
Started | 14 | 14 | 10 | 12
Completed | 14 | 13 | 8 | 11
Not Completed | 0 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Solicited Event | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose ChAd155-RG | High Dose ChAd155-RG (x1) | High Dose ChAd155-RG (x2) | RABAVERT | Total
Number analyzed (Participants) | 14 | 14 | 10 | 12 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (10.1) | 30.4 (8.6) | 28.6 (5.8) | 26.8 (4.4) | 29.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 7 | 9 | 33
  Male | 7 | 4 | 3 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 13 | 13 | 9 | 12 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 1 | 1 | 6
  White | 11 | 8 | 8 | 9 | 36
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 10 | 12 | 50
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.7 (4.3) | 27.5 (3.5) | 25.2 (3.6) | 26.5 (3.1) | 26.9 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Solicited Injection Site Reactogenicity Events in Each Treatment Arm and Overall
Description: Injection site reactogenicity events were solicited on a memory aid completed by participants from the time of each vaccination through Day 7 following each vaccination. Injection site reactogenicity events included pruritus, erythema, ecchymosis, induration/swelling, pain, and tenderness. Each event was graded as mild, moderate, or severe. Participants are counted according to their maximum severity of injection site event reported. Participants reporting no injection site events are counted under "None".
Time Frame: Day 1 through Day 29
Population: The Safety Population consists of all participants who received at least one dose of vaccine and for whom any data on safety are available.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants include every participant in the Low Dose ChAd155-RG arm, High Dose ChAd155-RG (x1) arm, High Dose ChAd155-RG (x2) arm, and RABAVERT arm.
Arm/Group | Low Dose ChAd155-RG | High Dose ChAd155-RG (x1) | High Dose ChAd155-RG (x2) | RABAVERT | All Participants
Number analyzed (Participants) | 14 | 14 | 10 | 12 | 50
Participants
  None | 3 | 2 | 0 | 0 | 5
  Mild | 10 | 11 | 8 | 9 | 38
  Moderate | 1 | 1 | 2 | 3 | 7
  Severe | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number and Percentage of Participants With Solicited Systemic Reactogenicity Events in Each Treatment Arm and Overall
Description: Systemic reactogenicity events were solicited on a memory aid completed by participants from the time of each vaccination through Day 7 following each vaccination. Systemic reactogenicity events included fever, chills/shivering/sweating, fatigue, malaise, myalgia and arthralgia (exclusive of the injection site), headache, and nausea. Each event was graded as mild, moderate, or severe. Participants are counted according to their maximum severity of systemic event reported. Participants reporting no systemic events are counted under "None".
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose ChAd155-RG | High Dose ChAd155-RG (x1) | High Dose ChAd155-RG (x2) | RABAVERT | All Participants
Number analyzed (Participants) | 14 | 14 | 10 | 12 | 50
Participants
  None | 3 | 1 | 1 | 4 | 9
  Mild | 5 | 4 | 3 | 3 | 15
  Moderate | 5 | 8 | 5 | 5 | 23
  Severe | 1 | 1 | 1 | 0 | 3

3. Primary Outcome: Number and Percentage of Participants With Serious Adverse Events (SAEs) Considered Study Vaccine-Related in Each Treatment Arm and Overall
Description: An AE or suspected AE was considered "serious" if, in the view of either the investigator or sponsor, it resulted in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
  Events were determined to be related if there was a reasonable possibility that the study product caused the AE; that is, there was evidence to suggest a causal relationship between the study product and the AE.
  Each event was graded as mild, moderate, or severe. Participants are counted according to their maximum severity of event reported. Participants reporting no vaccine-related SAEs are counted under "None".
Time Frame: Day 1 through Day 381
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose ChAd155-RG | High Dose ChAd155-RG (x1) | High Dose ChAd155-RG (x2) | RABAVERT | All Participants
Number analyzed (Participants) | 14 | 14 | 10 | 12 | 50
Participants
  None | 14 | 14 | 10 | 12 | 50
  Mild | 0 | 0 | 0 | 0 | 0
  Moderate | 0 | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number and Percentage of Participants With Study Vaccine-related Lab Adverse Events (AEs) in Each Treatment Arm and Overall
Description: Clinical safety lab parameters evaluated after receipt of vaccine (on Days 2, 8, 16, and Day 22) included WBCs, hemoglobin, platelets, absolute neutrophil count, absolute lymphocyte count, ALT, AST, total bilirubin, BUN, and creatinine. Lab events were assessed for relatedness and were determined to be related if there was a reasonable possibility that the study product caused the AE; that is, there was evidence to suggest a causal relationship between the study product and the AE.
  Each lab event was graded as mild, moderate, or severe. Participants are counted according to their maximum severity of event reported. Participants reporting no lab events are counted under "None".
Time Frame: Day 1 through Day 22
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose ChAd155-RG | High Dose ChAd155-RG (x1) | High Dose ChAd155-RG (x2) | RABAVERT | All Participants
Number analyzed (Participants) | 14 | 14 | 10 | 12 | 50
Participants
  None | 8 | 6 | 3 | 8 | 25
  Mild | 5 | 5 | 4 | 3 | 17
  Moderate | 1 | 3 | 2 | 1 | 7
  Severe | 0 | 0 | 1 | 0 | 1

5. Primary Outcome: Number and Percentage of Participants With Unsolicited Study Vaccine-related Adverse Events (AEs) in Each Treatment Arm and Overall
Description: Adverse events were defined as any untoward medical occurrence in a patient or clinical investigation participant administered a study product regardless of its causal relationship to the study product administration. Unsolicited, non-serious AEs were collected from participants from Day 1 through Day 28 after the last vaccination (Day 50).
  Events were determined to be related if there was a reasonable possibility that the study product caused the AE; that is, there was evidence to suggest a causal relationship between the study product and the AE.
  Each event was graded as mild, moderate, or severe. Participants are counted according to their maximum severity of event reported. Participants reporting no vaccine-related AEs are counted under "None".
Time Frame: Day 1 through Day 50
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose ChAd155-RG | High Dose ChAd155-RG (x1) | High Dose ChAd155-RG (x2) | RABAVERT | All Participants
Number analyzed (Participants) | 14 | 14 | 10 | 12 | 50
Participants
  None | 14 | 13 | 10 | 11 | 48
  Mild | 0 | 1 | 0 | 1 | 2
  Moderate | 0 | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number and Percentage of Participants With New Onset of a Chronic Medical Condition in Each Treatment Arm and Overall
Description: Participants were queried at each visit for the occurrence of new onset chronic medical conditions throughout the duration of the study.
Time Frame: Day 1 through Day 381
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose ChAd155-RG | High Dose ChAd155-RG (x1) | High Dose ChAd155-RG (x2) | RABAVERT | All Participants
Number analyzed (Participants) | 14 | 14 | 10 | 12 | 50
Participants | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number and Percentage of Participants With Serious Adverse Events (SAEs) in Each Treatment Arm and Overall
Description: An AE or suspected AE was considered "serious" if, in the view of either the investigator or sponsor, it resulted in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
  Each event was graded as mild, moderate, or severe. Participants are counted according to their maximum severity of event reported. Participants reporting no SAEs are counted under "None".
Time Frame: Day 1 through Day 381
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose ChAd155-RG | High Dose ChAd155-RG (x1) | High Dose ChAd155-RG (x2) | RABAVERT | All Participants
Number analyzed (Participants) | 14 | 14 | 10 | 12 | 50
Participants
  None | 14 | 14 | 10 | 12 | 50
  Mild | 0 | 0 | 0 | 0 | 0
  Moderate | 0 | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants Seroconverting to Rabies Virus in Each Treatment Arm and Overall
Description: Serum samples for rabies VNA were collected prior to vaccination (Day 1) and on Day 8, Day 15, Day 22, Day 29, Day 91, Day 181, and Day 381. Results from the rabies VNA RFFIT assay were reported in IU/mL, with a typical range of 1-15 IU/mL. Results beyond 15 IU/mL required dilution and retesting per the lab's standard operating procedures. The lower limit of quantification for the RFFIT assay is 0.1 IU/mL; values below the LLOQ were imputed as 1/2 the LLOQ, or 0.05 IU/mL. Seroconverting to rabies virus is defined as VNA concentration =0.5 IU/mL post-vaccination.
Time Frame: Day 8, Day 15, Day 22, Day 29, Day 91, Day 181, and Day 381
Population: The Modified Intent-to-Treat population consists of all subjects who received at least one dose of study vaccine and contributed both pre- and at least one post-study vaccination venous blood samples for immunogenicity testing for which valid results were reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Dose ChAd155-RG | High Dose ChAd155-RG (x1) | High Dose ChAd155-RG (x2) | RABAVERT | All Participants
Number analyzed (Participants) | 14 | 14 | 10 | 11 | 49
percentage of participants
  Day 8: number analyzed (Participants) | 13 | 14 | 10 | 11 | 48
  Day 8 | 0 [0 to 24.7] | 0 [0 to 23.2] | 0 [0 to 30.8] | 0 [0 to 28.5] | 0 [0 to 7.4]
  Day 15: number analyzed (Participants) | 14 | 14 | 9 | 11 | 48
  Day 15 | 43 [17.7 to 71.1] | 57 [28.9 to 82.3] | 89 [51.8 to 99.7] | 82 [48.2 to 97.7] | 65 [49.5 to 77.8]
  Day 22 | 50 [23 to 77] | 64 [35.1 to 87.2] | 100 [69.2 to 100] | 100 [71.5 to 100] | 76 [61.1 to 86.7]
  Day 29: number analyzed (Participants) | 14 | 13 | 9 | 11 | 47
  Day 29 | 64 [35.1 to 87.2] | 62 [31.6 to 86.1] | 100 [66.4 to 100] | 100 [71.5 to 100] | 79 [64.3 to 89.3]
  Day 91: number analyzed (Participants) | 10 | 10 | 6 | 8 | 34
  Day 91 | 40 [12.2 to 73.8] | 70 [34.8 to 93.3] | 67 [22.3 to 95.7] | 100 [63.1 to 100] | 68 [49.5 to 82.6]
  Day 181: number analyzed (Participants) | 14 | 10 | 9 | 11 | 44
  Day 181 | 29 [8.4 to 58.1] | 40 [12.2 to 73.8] | 33 [7.5 to 70.1] | 91 [58.7 to 99.8] | 48 [32.5 to 63.3]
  Day 381: number analyzed (Participants) | 14 | 9 | 8 | 8 | 39
  Day 381 | 29 [8.4 to 58.1] | 22 [2.8 to 60] | 13 [0.3 to 52.7] | 63 [24.5 to 91.5] | 31 [17 to 47.6]

9. Secondary Outcome: Rabies VNA Geometric Mean Titer
Description: Serum samples for rabies VNA were collected prior to vaccination (Day 1) and on Day 8, Day 15, Day 22, Day 29, Day 91, Day 181, and Day 381. Results from the rabies VNA RFFIT assay were reported in IU/mL, with a typical range of 1-15 IU/mL. Results beyond 15 IU/mL required dilution and retesting per the lab's standard operating procedures. The lower limit of quantification for the RFFIT assay is 0.1 IU/mL; values below the LLOQ were imputed as 1/2 the LLOQ, or 0.05 IU/mL. The geometric mean titer was calculated for each study arm at each immunogenicity time point.
Time Frame: Day 1, Day 8, Day 15, Day 22, Day 29, Day 91, Day 181, and Day 381
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Low Dose ChAd155-RG | High Dose ChAd155-RG (x1) | High Dose ChAd155-RG (x2) | RABAVERT | All Participants
Number analyzed (Participants) | 14 | 14 | 10 | 11 | 49
titer
  Day 1 | 0.05 [0.05 to 0.06] | 0.05 [NA to NA] — Not calculable due to insufficient variability. | 0.05 [NA to NA] — Not calculable due to insufficient variability. | 0.05 [NA to NA] — Not calculable due to insufficient variability. | 0.05 [0.05 to 0.05]
  Day 8: number analyzed (Participants) | 13 | 14 | 10 | 11 | 48
  Day 8 | 0.05 [0.05 to 0.06] | 0.05 [NA to NA] — Not calculable due to insufficient variability. | 0.05 [NA to NA] — Not calculable due to insufficient variability. | 0.06 [0.05 to 0.09] | 0.05 [0.05 to 0.06]
  Day 15: number analyzed (Participants) | 14 | 14 | 9 | 11 | 48
  Day 15 | 0.41 [0.15 to 1.16] | 0.54 [0.25 to 1.16] | 0.78 [0.44 to 1.38] | 0.89 [0.39 to 2.03] | 0.60 [0.40 to 0.89]
  Day 22 | 0.7 [0.28 to 1.76] | 0.79 [0.39 to 1.6] | 1.65 [0.86 to 3.17] | 2.35 [1.13 to 4.88] | 1.13 [0.78 to 1.66]
  Day 29: number analyzed (Participants) | 14 | 13 | 9 | 11 | 47
  Day 29 | 0.67 [0.27 to 1.65] | 0.68 [0.33 to 1.40] | 1.30 [0.73 to 2.31] | 10.58 [6.48 to 17.30] | 1.45 [0.91 to 2.33]
  Day 91: number analyzed (Participants) | 10 | 10 | 6 | 8 | 34
  Day 91 | 0.28 [0.10 to 0.80] | 0.49 [0.24 to 0.98] | 0.44 [0.20 to 0.96] | 2.49 [1.28 to 4.88] | 0.60 [0.38 to 0.95]
  Day 181: number analyzed (Participants) | 14 | 10 | 9 | 11 | 44
  Day 181 | 0.20 [0.08 to 0.50] | 0.37 [0.16 to 0.86] | 0.19 [0.10 to 0.37] | 0.92 [0.43 to 1.97] | 0.33 [0.22 to 0.51]
  Day 381: number analyzed (Participants) | 14 | 9 | 8 | 8 | 39
  Day 381 | 0.14 [0.06 to 0.31] | 0.16 [0.07 to 0.34] | 0.16 [0.07 to 0.34] | 0.84 [0.36 to 1.99] | 0.21 [0.14 to 0.33]

10. Secondary Outcome: Peak Rabies VNA Geometric Mean Titer
Description: Serum samples for rabies VNA were collected prior to vaccination (Day 1) and on Day 8, Day 15, Day 22, Day 29, Day 91, Day 181, and Day 381. Results from the rabies VNA RFFIT assay were reported in IU/mL, with a typical range of 1-15 IU/mL. Results beyond 15 IU/mL required dilution and retesting per the lab's standard operating procedures. The lower limit of quantification for the RFFIT assay is 0.1 IU/mL; values below the LLOQ were imputed as 1/2 the LLOQ, or 0.05 IU/mL. Peak geometric mean titer was defined for each study arm as the geometric mean of the highest titer per participant across all post-vaccination antibody timepoints.
Time Frame: Day 8 through Day 381
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Low Dose ChAd155-RG | High Dose ChAd155-RG (x1) | High Dose ChAd155-RG (x2) | RABAVERT | All Participants
Number analyzed (Participants) | 14 | 14 | 10 | 11 | 49
titer | 0.94 [0.37 to 2.36] | 0.90 [0.44 to 1.84] | 1.65 [0.86 to 3.17] | 10.63 [6.50 to 17.38] | 1.79 [1.15 to 2.79]

ADVERSE EVENTS:
Time Frame: Non-serious, unsolicited AEs were collected from Day 1 through Day 50. Serious adverse events and all-cause mortality were collected from Day 1 through Day 381.
Arm/Group | Low Dose ChAd155-RG | High Dose ChAd155-RG (x1) | High Dose ChAd155-RG (x2) | RABAVERT
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 13/14 | 14/14 | 10/10 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose ChAd155-RG (N=14) | High Dose ChAd155-RG (x1) (N=14) | High Dose ChAd155-RG (x2) (N=10) | RABAVERT (N=12)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (5) | 1 (1) | 3 (5) | 1 (1)
Fatigue (General disorders) | 8 (16) | 11 (16) | 9 (13) | 6 (8)
Feeling of body temperature change (General disorders) | 5 (6) | 6 (8) | 7 (8) | 3 (7)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 6 (7) | 10 (12) | 6 (8) | 4 (7)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 4 (4) | 3 (3)
Vaccination site erythema (General disorders) | 2 (3) | 2 (2) | 3 (5) | 3 (3)
Vaccination site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaccination site pain (General disorders) | 9 (19) | 11 (22) | 10 (29) | 11 (44)
Vaccination site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Blood urea increased (Investigations) | 0 (0) | 2 (6) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (4) | 1 (4) | 2 (6) | 3 (8)
Lymphocyte count decreased (Investigations) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 1 (8) | 1 (2) | 1 (1) | 2 (3)
White blood cell count decreased (Investigations) | 4 (6) | 4 (7) | 2 (2) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 1 (1) | 3 (5) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 9 (10) | 5 (10) | 4 (7)
Headache (Nervous system disorders) | 9 (17) | 13 (20) | 7 (13) | 5 (8)
Vulval disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT04019444/Prot_001.pdf
  • Statistical Analysis Plan (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT04019444/SAP_002.pdf
  • Informed Consent Form (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT04019444/ICF_000.pdf